CLINICAL TRIAL: NCT05652699
Title: High Flow Nasal Oxygen Therapy Re-evaluated from a Conceptual Point of View: Effect on Respiratory Effort and Lung Aeration After Extubation
Brief Title: Effect of HFNO Therapy on Respiratory Effort After Extubation
Acronym: T-REX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henrik Endeman (Other)
Collaborators: Franciscus Gasthuis (Other); Maasstad Hospital (Other)
Responsible Party: Sponsor-Investigator, Henrik Endeman, MD, PhD, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL80844.078.22
Record Dates: First submitted 2022-11-23; First posted 2022-12-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Failure; Post Extubation Acute Respiratory Failure Requiring Reintubation
Keywords: High-flow oxygen; Intensive Care Unit; Extubation; Reintubation; Respiratory Effort; Aeration
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Flow Nasal Oxygen (Active Comparator): 60L/minute. FiO2 according to clinical protocol. Temperature highest tolerated by patient, starting with 37 degrees Celcius.
  Interventions: Other: High Flow Nasal Oxygen
- Conventional Oxygen therapy (Active Comparator)
  Interventions: Other: Conventional Oxygen Therapy

INTERVENTIONS:
Other: High Flow Nasal Oxygen — Flow 60L/minute. FiO2 according to clinical protocol. Temperature highest tolerated by patient, starting with 37 degrees Celsius.
  Other Names: High Flow Nasal Cannula; Nasal High Flow Therapy
  Arms: High Flow Nasal Oxygen
Other: Conventional Oxygen Therapy — Nasal Cannula, Venturi Mask or Non-rebreathing mask, according to local clinical protocols
  Arms: Conventional Oxygen therapy

SUMMARY:
Rationale: Despite the lack of clear clinical protocols, High Flow Nasal Oxygen (HFNO) is used as post-extubation respiratory support. Although HFNO seems to reduce the need for re-intubation, scepticism on its use persists as the mechanism of action in post-extubation patients remains undefined. Monitoring weaning from invasive mechanical ventilation while monitoring respiratory effort might help to determine the added value of HFNO surrounding extubation. We hypothesize that HFNO, compared to conventional oxygen therapy (COT), prevents de-recruitment of the lung and reduces respiratory effort, and so provides a physiologic clarification for the reduction in the need for reintubation.

Objective: Determine the physiological effect of HFNO compared to COT in the extubation phase regarding respiratory effort and lung aeration.

Study design: A physiologic, randomized clinical study comparing two standard of clinical care therapies.

Study population: Adult patients on invasive mechanical ventilation (IMV) for >72 hours, who are scheduled for extubation.

Intervention (if applicable): Before extubation, patients are randomized to receive COT (reference group) or HFNO as oxygenation regimen after extubation.

Main study parameters/endpoints: The main outcome is the difference in change in lung respiratory muscle effort (mean ΔPES) at 24 hours post-extubation between the study groups. Secondary parameters are differences in changes in respiratory effort at 2 and 4 hours post-extubation, difference in change in lung aeration (mean ΔEELI), differences in tidal volume, dyspnea score, and respiratory and sputum parameters between patients undergoing different post-extubation oxygenation regimens.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Receiving IMV > 48 hours for any cause
* Successfully completing spontaneous breathing trial (SBT) as per local clinical guideline
* Provided written informed consent, through legal representatives on indication

Exclusion Criteria:

* Any clinical situation preventing appropriate execution of study procedures
* The presence of a tracheostomy
* Any feature that precludes HFNO-initiation
* Indication for NIV such as hypercapnia at end of SBT, or Obstructive/central Sleep Apnoea Syndrome or Obesity Hypoventilation Syndrome with CPAP use in medical history
* Contra-indication for nasogastric tube or inability to perform adequate PES measurements.
* Known diaphragm paralysis defined as elevated hemi-diaphragm on X-ray and evidence of paralysis during ultrasound (i.e. paradoxal diaphragm movement during sniffing)
* Known pregnancy or current breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
delta Esophageal Pressure (ΔPES) | At 24 hours after extubation
  The difference between groups in change in ΔPES in patients 24 hours post-extubation.

SECONDARY OUTCOMES:
ΔPES | At 2 and 4 hours post-extubation
  The difference between groups in change in ΔPES after extubation
delta global End-expiratory lung impedance (∆EELIglobal) | At 2, 4 and 24 hours after extubation
  Difference between the groups in change in mean ∆EELIglobal
Pressure-time product of Esophageal Pressure (PTPES) | At 2,4 and 24 hours after extubation
  The difference between the groups in mean pressure-time product (PTPES) compared to baseline.
EIT parameters | At 2, 4 and 24 hours after extubation
  ∆VARt, ∆EELIdependent, ∆EELInon-dependent compared to baseline (impedance on IMV).
Global Inhomogeneity index | At 2, 4 and 24 hours after extubation

OTHER OUTCOMES:
non-invasive positive pressure ventilation (NIPPV) | Within 7 days post-extubation
  Treatment escalation
Continuous positive airway pressure (CPAP) | Within 7 days post-extubation
  Treatment escalation
invasive mechanical ventilation (IMV). | Within 7 days post-extubation
  Treatment escalation
Survival rate | Within 7 days post-extubation
  Survival rates
Sputum | At 2 and 24 hours after extubation
  Difference in sputum aspect and sputum clearance between the study groups, assessed with a 5-point likert scale.
Dyspnea score | At 2 and 24 hours after extubation
  Difference in dyspnea sensation between the groups, measured with Visual Analog Scale (VAS, ranging from 0 = No dyspnea until 10 = maximum dyspnea).

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Janssen ML, Weller D, Wils EJ, Lupgens N, den Uil CA, Boer DP, Gommers DAMPJ, Heunks LMA, Jonkman AH, Endeman H. Physiological Effects of High-Flow Nasal Oxygen Compared With Conventional Oxygen Therapy: A Randomized Trial in Postextubation Patients. Crit Care Med. 2025 Dec 15. doi: 10.1097/CCM.0000000000006993. Online ahead of print. PMID 41395998